CLINICAL TRIAL: NCT03210857
Title: Effect of Voluntary Neck Extension in the Occurrence of an Increase in the Pulsatility Index of Right Internal Carotid Artery in the Amateur Diver, Performing an Apnoea of Two Minutes or More: a Prospective, Monocentric, Open Interventional Study
Brief Title: Effects of Voluntary Neck Extension on Cerebral Blood Flow, in Breath-hold Divers Ending an Apnoea of Two Minutes or More.
Acronym: APNECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC17_0163
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Healthy Amateur Divers
Keywords: apnea; neck extension; syncope; diving blackout; right internal carotid arteria; pulsatility index; healthy trained apnoea divers; doppler ultrasonography
MeSH Terms: conditions — Apnea; Syncope

STUDY DESIGN:
Intervention Model Description: Subject will realize an apnea of 2 minutes or more, depending on his abilities, and some parameters will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apnea performing (Experimental): The included subjects will make an apnea of two minutes or more, sitting on a chair with cold strips on the face, initially with the head in neutral position. Then, when they feel the end of their apnea, they will have to raise their left hand to signal it to the Doppler manipulator, who will then realize the apnea reference measurement.
  As soon as this is done, the subjects will be asked to perform an extension of the neck, so as to look at the ceiling. A final measurement will then be made in apnea, the head always in extension. Subjects then resume their breathing in this same position. A final measurement will then be made.
  Interventions: Other: apnea performing

INTERVENTIONS:
Other: apnea performing — The included subjects will make an apnea of two minutes or more, sitting on a chair with cold strips on the face, initially with the head in neutral position. Then, when they feel the end of their apnea, they will have to raise their left hand to signal it to the Doppler manipulator, who will then realize the apnea reference measurement.
  As soon as this is done, the subjects will be asked to perform an extension of the neck, so as to look at the ceiling. A final measurement will then be made in apnea, the head always in extension. Subjects then resume their breathing in this same position. A final measurement will then be made.

SUMMARY:
The aim of this study is to demonstrate the effect of the voluntary neck extension in the occurrence of an increase in the pulsatility index of the right internal carotid artery in the amateur diver, realizing an apnea of two minutes or more.

DETAILED DESCRIPTION:
In literature concerning apnoea, accidents have been described during neck extension.

Accidental drowning are frequent on the French coast every year and many of them concern apneists victims of apnoeic blackout.

Neck extension is thus suspected to possibly produce an apnoeic blackout at the end of the dive since 1965, when Sir Sciarli (diving medicine pioneer) suspected this hypothesis.

Physiologically, during a dive in apnea, the human cardiovascular system is subjected to a parasympathetic dominance, via the apnea reflex and the diving reflex. This parasympathetic dominant could be reinforced during a neck extension at the end of snorkeling during the ascent.

Hypothesis: the neck extension at the end of apnea contributes to increase the pulsatility index of the right internal carotid artery by vagal component and thus causes a decrease in cerebral blood flow and may lead to the initiation of syncope in the healthy amateur free diver or underwater fisherman.

ELIGIBILITY:
Inclusion Criteria:

* Major (≥18 years), under the age of 51
* Male
* Can hold an apnea of 2 minutes or more
* Practicing for less than 2 years the apnea at the rate of at least 10 sessions of apnea in the year
* Not having a known cardiovascular history : any form of heart rhythm disorder, Ischemic heart disease, angina, arteriopathy, any valvular pathology, high blood pressure ...
* No known respiratory history (asthma, Chronic Obstructive Pulmonary Disease, bronchiectasis, pulmonary emphysema, pneumothorax, pleurisy, pulmonary infection, lobectomy ...)
* No neurological history of type: epilepsy, deficit syndrome, iterative loss of knowledge, recent head trauma with loss of consciousness

Exclusion Criteria:

* - Minors and persons over 51 years of age
* Person under curators or trusteeship
* Person with a history of cardiovascular, respiratory or epilepsy as cited by the French Federation of Study and Submarine Sports, which poses as a contra-indication to the practice of apnea: Cardiac insufficiency, Obstructive Cardiomyopathy, syncopal risk pathology (valvulopathies type aorting narrowing or mitral narrowing), paroxysmal tachycardia, non-paired auriculo ventricular block 2/3, stroke, uncontrolled hypertension after stress test, recent infarction, angina, pericarditis. Asthma stage 3, severe Chronic Obstructive Pulmonary Disease, bronchiectasis, pulmonary emphysema, pneumothorax, pleurisy, pulmonary infection, lobectomy ...) Epilepsy, deficit syndrome, iterative loss of knowledge, recent head trauma with loss of consciousness in difficulty, symptomatic cervical or lumbar disc herniation
* Patient with medical treatment affecting the cardiovascular or respiratory system (for example: ventolin, betablocker ...)

Ages: 18 Years to 51 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Effect of the voluntary neck extension in the occurrence of an increase in the pulsatility index of the right internal carotid artery in the amateur diver, realizing an apnea of two minutes or more | 2 minutes or more: at the breaking point of apnea.
  To demonstrate the potential implication of cervical extension in the decrease of cerebral blood flow in amateur diver apnea by measuring the variation in the pulsatility index of the right internal carotid artery (RICAPI), by the intra-individual comparison of the RICAPI in amateur diver in rupture of apnea with neck extension (NE) versus the RICAPI of amateur diver in rupture of apnea without NE.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ANDRE, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes hospital, Nantes, France